CLINICAL TRIAL: NCT02944175
Title: Cerebral Oxygenation and Metabolism After Reversal Of Rocuronium Neuromuscular Blockade In Cases Of Supratentorial Tumors: A Comparative Study Between Sugammadex Versus Neostigmine
Brief Title: Cerebral Oxygenation and Metabolism After Reversal Of Rocuronium: Comparison Between Sugammadex Versus Neostigmine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MD ∕16.07.22
Record Dates: First submitted 2016-10-20; First posted 2016-10-25 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Supratentorial Brain Tumor Surgery
MeSH Terms: interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugammadex (Experimental): Patients will receive Sugammadex to antagonise the residual effects of neuromuscular blocking drugs
  Interventions: Drug: Sugammadex
- Neostigmine (Active Comparator): Patients will receive Neostigmine to antagonise the residual effects of neuromuscular blocking drugs
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex — At the end of surgery and when 2 responses were achieved on the TOF stimulation, Sugammadex 2 mg·kg-1 was administered intravenously in Group S
  Arms: Sugammadex
Drug: Neostigmine — At the end of surgery and when 2 responses were achieved on the TOF stimulation neostigmine 0.05 mg·kg-1 + atropine 0.02 mg·kg-1 was administered intravenously
  Arms: Neostigmine

SUMMARY:
Cholinesterase inhibitors such as Neostigmine and Edrophonium have been used to reverse neuromuscular blockade after surgery. However, these drugs have a relatively slow onset and have adverse effects associated with stimulation of muscarinic receptors. In addition, neostigmine cannot be used to reverse profound blockade.

Anesthetics may exert their effects on various facets of cerebral function such as cerebral metabolic rate (CMRO2), cerebral blood flow (CBF), cerebral blood flow-metabolism coupling, intra cranial pressure (ICP), autoregulation, vascular response to CO2 and brain electrical activity. The net result of all these effects of the anaesthetic agents combined with their systemic effects may prove beneficial or detrimental to an already diseased brain.

In neurosurgical patients, clear and rapid recovery is required to early assess the neurological status and to maintain the cerebral oxygenation and metabolism within the normal physiological values which may be saved by sugammadex.

DETAILED DESCRIPTION:
The aim of this study is to compare Sugammadex versus neostigmine as a reversal to the neuromuscular blockade of rocuronium in patients undergoing supratentorial tumors resection. Comparison will include hemodynamics, respiratory effort and degree of sedation.

Indicators of global cerebral oxygenation and haemodynamics will be calculated using jugular bulb and peripheral arterial blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical class status I - III .
* Patients scheduled for elective supratentorial brain tumor resection

Exclusion Criteria:

* Severe uncompensated cardiac disease.
* Severe uncompensated respiratory disease.
* Severe uncompensated hepatic disease.
* Severe uncompensated renal disease.
* Morbidly obese patients.
* Documented hypersensitivity to one of the used drugs.
* Surgery in sitting position
* Surgery in prone position
* Patients with altered level of consciousness.
* Pregnancy.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-09-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Time to recovery of the train-of-four (TOF) ratio to 0.9 | For 1 hour after surgery
  The time from start of administration of sugammadex or neostigmine to recovery of the train-of-four (TOF) ratio to 0.9

SECONDARY OUTCOMES:
Arterio-Jugular oxygen content difference | For 6 hours after the start of surgery
  Ca jO2 = CaO2-CjvO
Estimated cerebral metabolic rate for oxygen (eCMRO2) | For 6 hours after the start of surgery
  eCMRO2=Ca- jO2 x(PaCO2 ∕ 100) Where ……. Ca jO2 is arterio-jugular O2 content difference.
  * PaCO2 is arterial CO2 tension
Cerebral Extraction Rate of Oxygen (CEO2) | For 6 hours after the start of surgery
  Calculated as the differences between arterial and jugular bulb O2 saturations, CEO2 = SaO2 - SjvO2
Cerebral Blood Flow equivalent (CBFe) | For 6 hours after the start of surgery
  Which is an index of flow metabolism relationship, calculated as a reciprocal of arterio-jugular O2 content difference
Heart rate | For 6 hours after the start of surgery
Blood pressure | For 6 hours after the start of surgery
Central venous pressure | For 6 hours after the start of surgery
Peripheral oxygen saturation | For 6 hours after the start of surgery
End-tidal carbon dioxide tension | For 6 hours after the start of surgery
Sedation level | For 1 hour after extubation
Total dose of neuromuscular blockade used | For 6 hours after the start of surgery
Total dose of suggamadex or neostigmine used | For 30 min after the end of surgery
Cumulative opioids consumption | For 6 hours after the start of surgery
Recovery time (RT) | For 1 hour after surgery
  the time of restoration of neuromuscular conduction sufficient for extubation from stoppage of anaesthesia till the patient can obey commands
Time between administration of sugammadex or neostigmine to recovery | For 1 hour after surgery
  Time from start of administration of sugammadex or neostigmine to recovery of the train-of-four (TOF) ratio to 0.9

CONTACTS AND LOCATIONS:
Overall Officials: Sherif A Mousa, Study Chair — Department of Anaesthesia, Surgical Intensive Care and Pain Medicine, College of Medicine, Mansoura University, Mansoura, Egypt

IPD SHARING:
Plan to Share IPD: Undecided